CLINICAL TRIAL: NCT00963274
Title: Phase I Study of Bortezomib and Romidepsin in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma, Indolent B-Cell Lymphoma, Peripheral T-Cell Lymphoma or Cutaneous T-Cell Lymphoma
Brief Title: Bortezomib and Romidepsin in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12215; P30CA016059 (NIH); MCC-12215 (Other: VCU Massey Cancer Center); R21CA137823 (NIH); CDR0000652509 (Registry Identifier: PDQ)
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; hepatosplenic T-cell lymphoma; nodal marginal zone B-cell lymphoma; peripheral T-cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral | interventions — Bortezomib; romidepsin; Depsipeptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib + romidepsin (Experimental): Bortezomib via a short intravenous infusion (3-5 seconds) followed by romidepsin via a 4 hour intravenous infusion weekly x 3 every 4 weeks. In order to identify appropriate doses, different subjects will be treated with different drug doses and observed for the effects, especially the side effects associated with higher doses.
  Interventions: Drug: Bortezomib; Drug: Romidepsin

INTERVENTIONS:
Drug: Bortezomib — Starting dose: 1.3 mg/sq m
  Other Names: Velcade; PS-341
Drug: Romidepsin — Starting dose: 8 mg/sq m
  Other Names: depsipeptide; FK288

SUMMARY:
This phase I trial studies the side effects and best dose of giving bortezomib and romidepsin together in treating patients with chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), indolent B-cell lymphoma, peripheral T-cell lymphoma (PTCL) or cutaneous T-cell lymphoma (CTCL). Bortezomib and romidepsin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) for the combination of bortezomib and romidepsin administered weekly x 3 every (q) 4wk in patients with CLL/SLL, indolent B-cell lymphoma, PTCL or cutaneous T-cell lymphoma (CTCL).

Secondary

* Determine safety and tolerance and describe the toxicities of the combination.
* Demonstrate adequate methods for the assessment of pharmacodynamic responses of CLL cells to the combination with respect to effects on NF-kappa B (nuclear RelA and processing of p52 as a marker of p100 processing), expression of the NF-kappa B-dependent proteins XIAP and Bcl-xL, and Bim, and document pharmacodynamic responses observed in the course of this study * Document the pharmacodynamic responses associated with this regimen in these patients.
* Document the anticancer activity of this regimen in these patients.

OUTLINE: Patients receive bortezomib IV over 3-5 seconds and romidepsin IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples from patients with chronic lymphocytic leukemia are collected at baseline and after day 1 of course 1 of study treatment for pharmacodynamic and correlative laboratory studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

* CLL or SLL, relapsed or refractory
* Indolent B-cell lymphoma, relapsed or refractory:

  * Follicle center lymphoma, follicular or diffuse
  * Marginal zone B-cell lymphoma (splenic, nodal, extranodal [this includes mucosa associated lymphoid tissue (MALT)])
  * Lymphoplasmacytic lymphoma
* PTCL, relapsed or refractory:

  * Anaplastic large cell lymphoma, anaplastic lymphoma kinase (ALK)-positive
  * Anaplastic large cell lymphoma, ALK-negative
  * Angioimmunoblastic T-cell lymphoma
  * Enteropathy-associated T-cell lymphoma
  * Extranodal natural killer (NK)/T-cell lymphoma, nasal type
  * Hepatosplenic T-cell lymphoma
  * PTCL, not otherwise specified (NOS)
  * Subcutaneous panniculitis-like T-cell lymphoma
* CTCL:

  * CTCL with subtypes of mycosis fungoides Stage IB or higher, Sézary syndrome, or primary cutaneous anaplastic large cell lymphoma who have failed a previous systemic treatment, as per the following:
  * Stage IA plaque, IB, or IIA: At least 4 prior conventional and/or experimental regimens (topical or systemic, including psoralen-ultraviolet light [PUVA] and systemic corticosteroids)
  * Stage IIB, III, or IV: At least 1 prior systemic regimen (systemic corticosteroids alone or PUVA alone do not count as systemic regimens for this purpose) NOTE: Repeated use of the same regimen is considered 1 regimen
* Prior allogeneic stem cell transplant is allowed provided that all of the following conditions are met:

  * >= 6 months have elapsed since allogeneic transplant
  * No Graft vs. Host Disease (GVHD) is present
  * Not currently on immunosuppressive therapy
* No prior or concurrent CNS malignancy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC > 1,500/mm^3
* Platelet count > 75,000/mm^3
* Hemoglobin > 7.5 g/dL (transfusion allowed)
* Serum creatinine ≤ 1.2 mg/dL or actual or calculated creatinine clearance > 60 mL/min
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ ULN
* Serum potassium ≥ 3.5 mEq/L (supplementation allowed)
* Serum magnesium ≥ 1.7 mEq/L (supplementation allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* Willing and able to comply with protocol requirements
* No prior severe allergic reactions to bortezomib, boron, mannitol, or romidepsin
* No progressing toxicity secondary to bortezomib
* No grade 1 peripheral neuropathy with pain or ≥ grade 2 peripheral neuropathy by NCI-CTCAE criteria (v4.0) within the past 14 days
* No condition related to ischemic heart disease, heart failure, or the risk of torsades de pointes or sudden cardiac death, including any of the following:

  * History of sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes, or resuscitated cardiac arrest unless currently addressed with an implantable cardiac defibrillator
  * Baseline heart rate > 140 beats per minute
  * Known congenital long QT syndrome
  * QTc interval > 480 milliseconds
  * Type II second-degree atrio-ventricular (AV) block, third-degree AV block, or ventricular rate < 50 beats per minute
  * Myocardial infarction within the past 6 months

    * Patients who have had a myocardial infarction 6-12 months ago are eligible provided they are asymptomatic and have a negative cardiac risk assessment (i.e., treadmill stress test, nuclear medicine stress test, or stress echocardiogram)
  * Angina upon ordinary physical activity

    * Angina only with strenuous, rapid, or prolonged exertion allowed
  * ECG with evidence of cardiac ischemia, as defined by the following:

    * ST depression of ≥ 2 mm, measured from isoelectric line to ST segment
    * T-wave inversion ≥ 4 mm, measured from isoelectric line to peak of T-wave
  * NYHA class II-IV congestive heart failure
  * Known left ventricular ejection fraction < 40% by MUGA scan or < 50% by echocardiogram or MRI
  * Known hypertrophic cardiomegaly or restrictive cardiomyopathy
* No uncontrolled hypertension, defined as persistent blood pressure ≥ 160/95 mm Hg despite medical management
* No clinically significant active infection, including known HIV infection or hepatitis B or C
* No other malignancy within the past 3 years except completely resected basal cell carcinoma or squamous cell carcinoma of the skin, in situ malignancy, or curatively treated low-risk prostate cancer
* No concurrent medical condition that, in the investigator's opinion, would compromise study treatment or assessment of toxicity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy, radiation therapy or investigational agents. If steroids for cancer control have been used, patients must be off theses agents for at least 1 week before starting treatment. (Maintenance therapy for non-malignant disease with prednisone or steroid equivalent dose less than 10 mg/day is permitted)
* Prior allogeneic stem cell transplantation allowed provided all of the following conditions are met:
* Greater than or equal to 6 months have elapsed since allogeneic transplant
* No Graft vs. Host Disease (GVHD) is present
* More than 4 weeks since prior bortezomib
* No concurrent oral hormonal contraceptives
* No concurrent potent or moderate CYP3A4 inhibitors
* No concurrent anti-arrhythmic agents
* No concurrent treatment with any drugs that are generally accepted to having a risk of causing torsades de pointes (class 1 drugs)

  * Class 2 or 3 drugs allowed at the discretion of the investigator
* No other concurrent systemic therapy for the malignancy
* Concurrent warfarin (coumadin) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-04-26 (Actual); Primary Completion 2014-07-17 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 years
  Dose at which no more than 1 dose-limiting toxicity is observed in as many as 6 patients

SECONDARY OUTCOMES:
Pharmacodynamic responses | 2 years
  To explore candidate pharmacodynamic markers for use in subsequent phase II trials.

CONTACTS AND LOCATIONS:
Overall Officials: Beata Holkova, MD, Principal Investigator — Massey Cancer Center; Thomas C. Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Steven Grant, MD, Study Chair — Virginia Commonwealth University; Sho Ma, MD, PhD, Principal Investigator — Northwestern University & Robert H Lurie Comprehensive Cancer Center; Amy Kimball, MD, PhD, Principal Investigator — University of Maryland Greenebaum Cancer Center; Nishitha Reddy, MBBS, Principal Investigator — Vanderbilt-Ingram Cancer Center, Vanderbilt University
Locations (5):
- United States (5):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Vanderbilt University, Nashville, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Holkova B, Yazbeck V, Kmieciak M, Bose P, Ma S, Kimball A, Tombes MB, Shrader E, Wan W, Weir-Wiggins C, Singh A, Hogan KT, Conine S, Sankala H, Roberts JD, Shea TC, Grant S. A phase 1 study of bortezomib and romidepsin in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma, indolent B-cell lymphoma, peripheral T-cell lymphoma, or cutaneous T-cell lymphoma. Leuk Lymphoma. 2017 Jun;58(6):1349-1357. doi: 10.1080/10428194.2016.1276287. Epub 2017 Jan 19. PMID 28103725
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/